CLINICAL TRIAL: NCT04119414
Title: Increasing Early Infant Male Circumcision Uptake in Zambia: Like Father Like Son
Brief Title: Like Father Like Son
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen Weiss, Research Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20190354; R34MH121111 (NIH)
Record Dates: First submitted 2019-10-06; First posted 2019-10-08 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Health Knowledge, Attitudes, Practice; Health Risk Behaviors
Keywords: Early Infant Male Circumcision; HIV infection
MeSH Terms: conditions — Behavior; Health Risk Behaviors; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S&S + LFLS Group (Experimental): 300 expecting couples totaling 600 participants will be completing the S&S program followed by the LFLS Program.
  Interventions: Behavioral: Spear and Shield (S&S) Program; Behavioral: Like Father Like Son (LFLS) Program

INTERVENTIONS:
Behavioral: Spear and Shield (S&S) Program — The S&S Program is a comprehensive sexual risk reduction intervention consisting of 4 weekly 90-minute manualized group sessions conducted by a trained Community Health Center (CHC) facilitator.
Behavioral: Like Father Like Son (LFLS) Program — The LFLS Program is a private 2 90-minute session conducted by a trained CHC facilitator. The sessions will be focused on exploring issues relevant to parental decision making related to voluntary medical male circumcision (VMMC) and early infant male circumcision (EIMC). Session 1 will be conducted antenatal and Session 2 will be immediately post-partum.

SUMMARY:
This purpose of this study is to look at the best way to offer the Like Father Like Son + Spear & Shield program.

ELIGIBILITY:
Inclusion Criteria:

* Men and women must be able to understand and sign the Informed Consent in English or local language.
* All participants must be adults able to provide consent
* Women participants may be pregnant
* Individuals not yet adults (infants, children, teenagers) are not eligible to participate
* Prisoners will not be eligible for recruitment

Exclusion Criteria:

- Participants not meeting any of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Weiss, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Lusaka Province Community Health Clinics, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The pilot study randomized 8 clinics to Experimental and Observation conditions. Participants were recruited from the four Experimental clinics. All expecting parents received the S&S + LFLS intervention. However, the circumcision outcomes were ultimately only measured in male infant and male adult participants.
  Observation clinics were not intended to recruit participants and as such, only clinic level data was intended to be obtained. These clinics ultimately did not provide their data.
Units Other Than Participants: Clinics
Groups:
- S&S + LFLS Group: 300 expecting couples totaling 600 participants will be completing S&S + LFLS, in 4 different clinics.
  Spear and Shield (S&S) Program: The S&S Program is a comprehensive sexual risk reduction intervention consisting of 4 weekly 90-minute manualized group sessions conducted by a trained Community Health Center (CHC) facilitator.
  Like Father Like Son (LFLS) Program: The LFLS Program is a private 2 90-minute session conducted by a trained CHC facilitator. The sessions will be focused on exploring issues relevant to parental decision making related to voluntary medical male circumcision (VMMC) and early infant male circumcision (EIMC). Session 1 will be conducted antenatal and Session 2 will be immediately post-partum.
Period: Overall Study
Arm/Group | S&S + LFLS Group
Started | 600; 8 Clinics
Completed | 300; 4 Clinics
Not Completed | 300; 4 Clinics
Not completed — 300 couples did not have a male child, and 4 clinics were only observed | 300

BASELINE CHARACTERISTICS:
Arm/Group | S&S + LFLS Group
Number analyzed (Participants) | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.53 (7.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300
  Male | 300
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 600
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Zambia | 600

OUTCOME MEASURES:

1. Primary Outcome: Number of Early Infant Male Circumcision
Description: As measured by the number of male infants who received circumcision during the first 60 days of life
Time Frame: Up to 60 days of life
Measure: Number; unit: participants
Groups:
- S&S + LFLS Group: 300 expecting couples totaling 600 participants will be completing the S&S program followed by the LFLS Program, in 4 different clinics.
  Spear and Shield (S&S) Program: The S&S Program is a comprehensive sexual risk reduction intervention consisting of 4 weekly 90-minute manualized group sessions conducted by a trained Community Health Center (CHC) facilitator.
  Like Father Like Son (LFLS) Program: The LFLS Program is a private 2 90-minute session conducted by a trained CHC facilitator. The sessions will be focused on exploring issues relevant to parental decision making related to voluntary medical male circumcision (VMMC) and early infant male circumcision (EIMC). Session 1 will be conducted antenatal and Session 2 will be immediately post-partum.
Arm/Group | S&S + LFLS Group
Number analyzed (Participants) | 600
participants | 300

2. Primary Outcome: Number of Voluntary Medical Male Circumcision
Description: Number of Voluntary Medical Male Circumcision (VMMC) of adult male participants within the total number of clinic patients being seen at each of the participating clinics.
Time Frame: Up to 12 months
Measure: Number; unit: participants
Groups:
- S&S + LFLS Program: 300 expecting couples totaling 600 participants will be completing the S&S program followed by the LFLS Program, in 4 different clinics.
  Spear and Shield (S&S) Program: The S&S Program is a comprehensive sexual risk reduction intervention consisting of 4 weekly 90-minute manualized group sessions conducted by a trained Community Health Center (CHC) facilitator.
  Like Father Like Son (LFLS) Program: The LFLS Program is a private 2 90-minute session conducted by a trained CHC facilitator. The sessions will be focused on exploring issues relevant to parental decision making related to voluntary medical male circumcision (VMMC) and early infant male circumcision (EIMC). Session 1 will be conducted antenatal and Session 2 will be immediately post-partum.
Arm/Group | S&S + LFLS Program
Number analyzed (Participants) | 300
participants | 150

3. Primary Outcome: Number of Parents' Who Indicate They Plan to Circumcise Their Infants
Description: Number of parents who indicate they plan to circumcise their infants prior to infants being born.
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | S&S + LFLS Program
Number analyzed (Participants) | 600
participants | 324

4. Primary Outcome: Clinic Level (Cluster) Number of Early Infant Male Circumcision (EIMC)
Description: Clinic Level (Cluster) Number of EIMC within the total number of clinic patients being seen at each of the participating clinics
Time Frame: 30 months
Population: Participating clinics did not provide data that included the number of EIMCs for analysis.
Arm/Group | S&S + LFLS Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | S&S + LFLS Group
All-Cause Mortality (participants affected / at risk) | 0/600
Serious Adverse Events (participants affected / at risk) | 0/600
Other Adverse Events (participants affected / at risk) | 0/600

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT04119414/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT04119414/ICF_002.pdf